CLINICAL TRIAL: NCT04574063
Title: Pilot of Lifestyle InterventiON to reducE brEast Cancer RiSk (PIONEER)
Brief Title: PIONEER Study of Lifestyle Intervention to Reduced Breast Cancer Risk
Acronym: PIONEER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCR 5113
Record Dates: First submitted 2020-09-07; First posted 2020-10-05 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Lifestyle Risk Reduction
MeSH Terms: conditions — Breast Neoplasms; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Breast cancer risk leaflet only (No Intervention)
- Breast cancer risk leaflet PLUS SNPs (No Intervention)
- Lifestyle website only (Experimental)
  Interventions: Behavioral: Lifestyle intervention to reduce breast cancer risk
- Lifestyle website PLUS SNPs (Experimental)
  Interventions: Behavioral: Lifestyle intervention to reduce breast cancer risk
- Lifestyle website PLUS group coaching (Experimental)
  Interventions: Behavioral: Lifestyle intervention to reduce breast cancer risk
- Lifestyle website PLUS group coaching PLUS SNPs (Experimental)
  Interventions: Behavioral: Lifestyle intervention to reduce breast cancer risk

INTERVENTIONS:
Behavioral: Lifestyle intervention to reduce breast cancer risk — Women will be educated about lifestyle factors which increase breast cancer risk. They will also be guided through an online goal setting process.
  Arms: Lifestyle website PLUS SNPs; Lifestyle website PLUS group coaching; Lifestyle website PLUS group coaching PLUS SNPs; Lifestyle website only

SUMMARY:
A randomised controlled trial in which women discharged from the symptomatic breast clinic, who are above population risk (according to Tyrer Cuzick) will be asked to create lifestyle related goals. They will be told their estimated risk of developing breast cancer and will be randomised to one of three interventions:

* Breast cancer risk leaflet only
* lifestyle website
* lifestyle website plus group coaching.

Fifty per cent of women will also be randomised to have Single Nucleotide Polymorphisms (SNPs) performed, and these will be incorporated into their risk score.

The primary end point will be whether or not women achieve their lifestyle goal.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged between 30 and 60 years
* Attending the symptomatic breast clinic at RMH Sutton or Chelsea OR the family history clinics at RMH Sutton or Chelsea, or has heard about the study through other means such as (but not limited to), friends who have been diagnosed with cancer, friends who are already taking part in the PIONEER study, social media, mainstream media, fliers through the doors of houses in the area of RMH.
* Benign or B3 diagnosis if participant has attended clinic
* Agree to receive their personalised breast cancer risk
* Available to participate in a 1 year risk prevention programme
* Able to attend the Royal Marsden for a blood test if randomised to this group

Exclusion Criteria:

* Malignant Diagnosis
* Does not want to find out personalised breast cancer risk
* Not available to participate for the full year
* NOTE: after risk assessment, women who have a breast cancer risk lower than that of population level will be excluded from participating in the behavioural change elements.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Goal achievement | Women will be asked this 12 months after entering the study
  Whether women have achieved their lifestyle goals. Proportion answering "yes" to a binary question: Did you achieve the goal you set? Compared between the three arms.

SECONDARY OUTCOMES:
To assess the acceptability of women to find out their personalised breast cancer risk and to commit to making a change in a modifiable risk factor | Measured when recruitment is complete, estimated at 3 months from start date
  Proportion of women approached who go on to join the study
To assess the acceptability of randomisation to different arms of intervention | Measured when the final participant has completed 12 months in the study, estimated 15 months from start date
  Attrition rate after randomisation within each group
To assess the impact of SNP testing on changes in behavioural risk factors | Measured when the final participant has completed 12 months in the study estimated 15 months from start date
  Goal achievement in SNP group compared with goal achievement in non-SNP group.
To assess the impact of the different interventions on changes in behavioural risk factors | Measured when the final participant has completed 12 months in the study estimated 15 months from start date
  Goal achievement compared between leaflet only group, website group and website + coaching group.
To assess the impact of knowledge of breast cancer risk on cancer anxiety scores | Measured when the final participant has completed 12 months in the study estimated 15 months from start date
  Change in Cancer Worry Scale (Revised) score from 0 to 3 months. Cancer Worry score is measured between 8 and 32 with 32 being the highest level of anxiety.
To identify whether there is an association between initial Cancer Worry Scale (Revised) score and change in behavioural risk factors | Measured when the final participant has completed 12 months in the study estimated 15 months from start date
  Cancer Worry score compared with goal achievement. Cancer Worry score is between 8 and 32 with 32 being the highest level of anxiety.
To identify whether commitment to a study of this design is sustainable and affected by study group | Measured when the final participant has completed 12 months in the study estimated 15 months from start date
  Participant retention rate.
To assess the impact of the different interventions on uptake and adherence to chemoprevention at 1 year | Measured when the final participant has completed 12 months in the study estimated 15 months from start date
  Proportion of women still taking chemoprevention at close of study compared between the three arms.
To consider the scalability of each element of the pilot study | Measured when the final participant has completed 12 months in the study estimated 15 months from start date
  Administration time required for each group; Average goal achievement compared to average cost of each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rusby, Principal Investigator — The Royal Marsden Hospital
Locations (1):
- The Royal Marsden Hospital NHS Foundation Trust, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Law R, Krupa K, Rusby J. Preventative therapy for breast cancer: a clinical experience. Breast Cancer Res Treat. 2023 Sep;201(2):205-213. doi: 10.1007/s10549-023-06985-1. Epub 2023 Jun 19. PMID 37336835